CLINICAL TRIAL: NCT01175733
Title: Chemoradiation With Gemcitabine in Combination With Panitumumab for Patients With Locally Advanced Pancreatic Cancer
Acronym: Vectibix
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, H.M.W. Verheul, Prof. Dr., Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080686
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Pancreatic Cancer
Keywords: Panitumumab; Chemoradiation; Pancreatic cancer; Locally advanced; Inoperable
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab (Experimental)
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — During the first 6 weeks Panitumumab will be administered weekly in combination with radiotherapy plus gemcitabine. From week 8 and further gemcitabine will be administered as monotherapy until disease progression or unacceptable toxicity, for a maximum duration of 1 year.

SUMMARY:
The purpose of this study is to investigate whether the addition of panitumumab to radiotherapy plus gemcitabine will increase the number of patients who are alive and progression free at 7 months.

DETAILED DESCRIPTION:
This is a phase I/II, multi-center dose escalation study.

Phase I:

Patients will be enrolled in cohorts of 3 per dose level until the MTD of panitumumab has been established.

Phase II:

Up to approximately 56 patients will be treated at the MTD level of panitumumab as established in the phase I part of the study.

Based on the historic data of patients with pancreatic cancer treated with gemcitabine based chemoradiation, we aim to increase the number of patients who are alive and progression free at 7 months from the historical value of 50% to 70% with the combination treatment of chemoradiation plus panitumumab.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed pancreatic cancer.
* Not eligible for curative resection.
* No distant metastases present.
* Previously untreated with chemotherapy and anti-cancer biologicals for current malignancy.
* No other current malignant disease, except for basal cell carcinoma of the skin.
* Measurable or evaluable disease as defined by RECIST 1.1 criteria.
* Performance status 0-2 Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) Scale.
* Age ≥ 18 years.
* Adequate haematological and biological functions:

  * Bone marrow function:

    1. Neutrophils ≥ 1.5 x 109/L
    2. Platelets ≥ 100 x 109/L
    3. Hb ≥ 6 mmol/L
  * Hepatic function:

    1. AST/ALT and alkaline phosphatase (ALP) ≤ 2.5 x institutional upper limit of normal (ULN)
    2. Bilirubin ≤ 1.5 times institutional ULN
  * Renal function:

eGFR >50ml/min

• Metabolic Function:

1. Magnesium ≥ lower limit of normal
2. Calcium ≥ lower limit of normal.

   * No imminent bowel obstruction.
   * No active bleeding.
   * No uncontrolled infection.
   * Patients with reproductive potential must use effective contraception. Female patients must have a negative pregnancy test.
   * Signed informed consent.

Exclusion Criteria:

* Participation in another therapeutic clinical study within 30 days of enrollment or during this clinical study.
* No adequate radiation therapy possible: based on the opinion of the radiation oncologist when radiation therapy cannot be performed because radiation field is too large (PTV volume too large or OAR too high)
* History of allergic reactions to gemcitabine or antibody treatment.
* Presence of any serious concomitant systemic disorders incompatible with the clinical study (e.g. uncontrolled inter-current illness including ongoing or active infection, uncontrolled hypertension).
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) within 1 year before enrolment/randomization
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan
* Presence of any significant central nervous system or psychiatric disorder(s) that would hamper the patient's compliance.
* Pregnant or breastfeeding women.
* Absence of adequate contraception for both male and female fertile patients for the duration of the study; and also for six months after last treatment.
* Known positive status for HIV and/or hepatitis B or C.
* Any reason why, in the investigator's opinion, the patient should not participate in the study.
* Drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07-08 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Phase I: the recommended safe dosing for the combination of chemoradiation with gemcitabine plus panitumumab. | 43 days
  During the phase I part of the study, we have planned to study four dose levels of panitumumab if no MTD is being derived before the final dose level. Patients will be enrolled in cohorts of 3 per dose level. If there are no dose-limiting toxicities (DLTs) experienced by the first 3 patients in a cohort during the first 43 days after the first study treatment, additional patients will be entered in the next dose level. At the final dose level recommended for the phase II study a minimum of 6 patients will be treated.
Phase II: the proportion of patients that is alive and progression-free at 7 months. | 1 year
  For each patient, the time of progression will be recorded. Any patient who discontinues treatment due to adverse reactions, refusal, or who goes on to receive alternate therapy will be considered censored at their last tumor assessment. The sample size was determined based upon a Bryant Day Phase II clinical trial design, taking into account both activity as well as toxicity. The proportion of patients with 7 month PFS will be calculated with exact 95% confidence intervals.
Phase II: safety and tolerability | 1 year
  Toxicities will be tabulated and summarized overall and across grade and type according to CTC criteria. When grade ≥3 toxicity occurs in ≥ 50% of patients this will be evaluated as unacceptable toxicity according to the two step evaluation design as described. This relatively high percentage of toxicity is based on the details of multiple studies of combination chemoradiation with gemcitabine as given in the introduction.

SECONDARY OUTCOMES:
Early signs of clinical activity of the combination of chemoradiation with gemcitabine plus panitumumab. | 1 year
  The assessment of early signs of clinical activity will be determined based upon CT-scan evaluation, pain relieve and decay in CA19.9 (where applicable).
Clinical response rate of the combination of chemoradiation with gemcitabine plus panitumumab. | 1 year
  The response rate will be determined as the proportion of treated patients who had a partial or complete response (as defined in Response Criteria section).
Time-to-progression (TTP) and overall survival | 1 year
  TTP and overall survival will be described in all patients using Kaplan-Meier curves. TTP will be defined based on CT-scan imaging based on Response Criteria according to RECIST (version 1.1) preferably or based on clinical evaluation and will be measured from enrolment. In addition, analyses of TTP will include death as being progressive disease. Kaplan-Meier curves will be used to summarize the pattern of TTP and overall survival. M median TTP and overall survival will be calculated along with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Henk MW Verheul, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands